CLINICAL TRIAL: NCT02190084
Title: Repetitive Transcranial Magnetic Stimulation for Apathy in Alzheimer's Dementia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Central Arkansas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Prasad R. Padala, Associate Director for clinical programs, GRECC, Central Arkansas Veterans Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 547461
Record Dates: First submitted 2014-07-11; First posted 2014-07-15 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Apathy; Alzheimer's Dementia
Keywords: apathy; Alzheimer's; executive function
MeSH Terms: conditions — Lethargy; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- transcranial magnetic stimulator (Active Comparator): Neurostar repetitive transcranial magnetic stimulator. The active procedure will stimulate at 120% motor threshold for 4 seconds at a frequency of 10 Hz, with an inter-train interval of 26 seconds for a total of 3,000 pulses. 20 treatment sessions are given over a four week period.
  Interventions: Device: Neurostar repetitive transcranial magnetic stimulator
- Sham coil treatment (Sham Comparator): Neurostar repetitive transcranial magnetic stimulator. 20 treatments identical in duration will be administered over a four week period.
  Interventions: Device: Neurostar repetitive transcranial magnetic stimulator

INTERVENTIONS:
Device: Neurostar repetitive transcranial magnetic stimulator — The active procedure will stimulate at 120% motor threshold for 4 seconds at a frequency of 10 Hz, with an inter-train interval of 26 seconds for a total of 3,000 pulses. 20 treatment sessions are given over a four week period.
  Other Names: •rTMS

SUMMARY:
Alzheimer's Dementia (AD) is a major public health problem. Apathy, a profound loss of motivation, is seen in majority of patients with AD. Dysfunction of the front of the brain and loss of dopamine, a type of neurochemical, in this part of brain results in apathy. Presence of apathy is linked to deficits in planning sequential tasks such as keeping a routine. Patients with apathy have poor physical function and their caregivers experience extra burden. Unfortunately there are no good medications to treat apathy. FDA has approved the use of brain stimulation by a magnet known as repetitive transcranial magnetic stimulation (rTMS), for treatment of depression. rTMS increases dopamine when applied to frontal lobe of brain so we propose that rTMS would be a good treatment option for apathy in AD. Study hypotheses include that rTMS to the dorsolateral prefrontal cortex (DLPFC) will improve apathy and executive function better than sham treatment in those with AD.

DETAILED DESCRIPTION:
Objective: Alzheimer's Dementia (AD) is a major public health problem. Apathy, a profound loss of motivation, is seen in majority of patients with AD. Dysfunction of the front of the brain and loss of dopamine, a type of neurochemical, in this part of brain results in apathy. Presence of apathy is linked to deficits in planning sequential tasks such as keeping a routine. Patients with apathy have poor physical function and their caregivers experience extra burden. Unfortunately there are no good medications to treat apathy. FDA has approved the use of brain stimulation by a magnet known as repetitive transcranial magnetic stimulation (rTMS), for treatment of depression. rTMS increases dopamine when applied to frontal lobe of brain so we propose that rTMS would be a good treatment option for apathy in AD.

Specific Aims: To determine the efficacy of rTMS to the dorsolateral prefrontal cortex (DLPFC) in treating apathy in mild AD in comparison to sham treatment.

• To compare the efficacy of rTMS to the DLPFC on executive function in mild AD in comparison to sham treatment.

Research Plan: Current study is a prospective randomized sham controlled study of daily rTMS.

Methods: Up to 500 subjects will be pre-screened to enroll 100 subjects for screening and randomizing up to 50 subjects to analyze 20 completers. Subjects with mild AD and apathy will be randomly assigned to rTMS or sham treatment after consent. All subjects will be tested for memory, behavioral problems, functioning and caregiver burden. Apathy will be assessed using the Apathy Evaluation Scale. Memory, executive function, functional status and caregiver burden will be assessed. Subjects will receive daily treatments for 4 weeks with either rTMS or sham coil for a total of 20 treatments. Neither the subject nor the investigators will know which treatment the subject is receiving. Testing will be repeated at the end of 4 weeks and at 8 and 12 weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age ≥ 55 years,
2. Diagnosis of Alzheimer's dementia meeting the DSM-IV TR criteria,
3. Apathy Evaluation Scale-Clinician (AES-C) score of ≥ 30,
4. Mini Mental Status Examination (MMSE) ≥ 18,
5. Subjects who clear the TMS adult safety scale (TASS)
6. On stable dose of antidepressants or dementia medicines (if applicable) for at least two months

Exclusion Criteria:

1. Subjects taking medications known to increase the risk of seizures from the 2012 Beers criteria: Bupropion, chlorpromazine, clozapine, maprotiline, olanzapine, thioridazine, thiothixene, and tramadol.
2. Subjects taking medications known to increase seizure threshold not listed in the Beers criteria but in the opinion of PI increase seizure threshold: tricyclic antidepressants, theophylline, methylphenidate, and high-dose thyroid supplementation.
3. Subjects taking ototoxic medications: Aminoglycosides, Cisplatin.
4. Subjects in current episode of major depression
5. History of bipolar disorder
6. Subjects with history of seizure or first degree relative with seizure disorder
7. Subjects with implanted device: wearable or implantable cardioverter defibrillators, conductive, ferromagnetic, or other magnetic sensitive metals that are implanted or are non-removable within 30 cm of the treatment coil or those with cochlear implants
8. Subjects with diagnosis of current alcohol related problems
9. Subjects with history of stroke , aneurysm, or cranial neurosurgery
10. Any condition that in the opinion of the study physician is likely to compromise their ability to safely participate in the study

Ages: 55 Years to 91 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Apathy Evaluation Scale (AES) | 4 weeks
  AES is an 18-item scale that assesses apathy in behavioral, cognitive and emotional domains over the previous four weeks.

SECONDARY OUTCOMES:
Trials making test | 4 weeks
  Widely used test for assessment of executive function.

OTHER OUTCOMES:
Exit 25 | 4 weeks
  EXIT-25 is a bedside measure of executive function. It defines the behavioral sequelae of executive dyscontrol and provides a standardized clinical encounter in which they can be observed.

CONTACTS AND LOCATIONS:
Locations (1):
- Central Arkansas Veterans Healthcare System, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Padala PR, Boozer EM, Lensing SY, Parkes CM, Hunter CR, Dennis RA, Caceda R, Padala KP. Neuromodulation for Apathy in Alzheimer's Disease: A Double-Blind, Randomized, Sham-Controlled Pilot Study. J Alzheimers Dis. 2020;77(4):1483-1493. doi: 10.3233/JAD-200640. PMID 32925060